CLINICAL TRIAL: NCT05596695
Title: The Effect of Minimizing Blood Pressure Variability on Postoperative Nausea and Vomiting in Women Undergoing Non-cardiac Surgery With Minor to Moderate Risk - a Prospective Randomized Clinical Trial
Brief Title: Minimisation of Blood Pressure Variability and Postoperative Nausea and Vomiting
Acronym: SICK
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Christian Reiterer, Principal Investigator, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: SICK_01
Record Dates: First submitted 2022-10-24; First posted 2022-10-27 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-07

CONDITIONS: PONV; Blood Pressure; Postoperative Recovery
Keywords: Blood Pressure Variability; Minor- to moderate-risk noncardiac surgery
MeSH Terms: conditions — Postoperative Nausea and Vomiting

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Intraoperative blood pressure management will be performed to maintain a systolic blood pressure of 120 ±5mmHg using a continuous infusion of a vasopressor starting at induction of anesthesia.
  Interventions: Other: Minimizing blood pressure variability
- Standard of Care Group (No Intervention): Intraoperative blood pressure management will be performed according to local clinical standard of care.

INTERVENTIONS:
Other: Minimizing blood pressure variability — Intraoperative blood pressure management will be performed to maintain a systolic blood pressure of 120 ±5mmHg using a continuous infusion of a vasopressor starting at induction of anaesthesia.
  Arms: Intervention Group

SUMMARY:
Intraoperative hypotension is associated with postoperative nausea and vomiting (PONV). Even though the exact mechanism linking PONV and hypotension is still unclear, a reduced intestinal tissue perfusion might trigger nausea and vomiting. Still to date only limited data evaluating intraoperative blood pressure and the incidence of PONV after general anesthesia exits. Furthermore, the effect of intraoperative blood pressure variability on the incidence of PONV has not been investigated yet. Therefore, we will test our primary hypothesis that the incidence of PONV during the early (0-2h) postoperative period will be minimized by targeting intraoperative blood pressure variability to a SPB of 120±5mmHg by using a continuous vasopressor infusion in female patients undergoing elective minor to moderate risk non-cardiac surgery.

DETAILED DESCRIPTION:
Background: Intraoperative hypotension is associated with postoperative nausea and vomiting (PONV). Even though the exact mechanism linking PONV and hypotension is still unclear, a reduced intestinal tissue perfusion might trigger nausea and vomiting. Still to date only limited data evaluating intraoperative blood pressure and the incidence of PONV after general anesthesia exits. Furthermore, the effect of intraoperative blood pressure variability on the incidence of PONV has not been investigated yet. Therefore, we will test our primary hypothesis that the incidence of PONV during the early (0-2h) postoperative period will be minimized by targeting intraoperative blood pressure variability to a SPB of 120±5mmHg by using a continuous vasopressor infusion in female patients undergoing elective minor to moderate risk non-cardiac surgery.

Methods: We will include 272 women between 18 and 50 years of age undergoing minor- to moderate-risk noncardiac surgery in this randomized, double-blinded clinical trial. Patients will randomly be assigned to intraoperative management of blood pressure with a SPB of 120±5mmHg (intervention group) or standard of care intraoperative blood pressure management (control group). Our primary outcome will be the incidence of PONV during the early (0-2h) postoperative period between the groups. Nausea will be assessed in 15-min intervals in the PACU for the first two postoperative hours on a 100mm visual analog scale. A PONV episode will be defined as the occurrence of nausea (VAS 50mm or greater) or vomiting.

Statistics: The primary outcome, the incidence of PONV during the early (0-2 hours) postoperative period will be compared between the intervention and control group using a Chi- Square-Test.

Level of originality: Data regarding the effects of intraoperative blood pressure on PONV are very limited and mainly available from retrospective analysis. So far, the effects of blood pressure variability on PONV have not been investigated yet. As PONV is still one of the most common complications after general anaesthesia leading to delayed discharge from PACU, patient discomfort and increased medical costs, it is important to search for additional methods to manage PONV. Our patient population, being at increased risk of PONV, could therefore profit from a more rapid postoperative recovery.

ELIGIBILITY:
Inclusion Criteria:

* Women 18-50 years of age at time of surgery
* ASA physical status I and II
* Scheduled for elective minor or moderate risk non-cardiac surgery with expected time of surgery ≥1 hour

Exclusion Criteria:

* Patients undergoing emergency surgery
* Scheduled for pheochromocytoma surgery
* Nausea and/or vomiting on the morning before surgery
* Taking anti-emetic drugs
* Pregnancy
* Dysfunction of the vestibular system

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 272 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
PONV | First two postoperative hours
  Incidence of postoperative nausea and vomiting within the first two postoperative hours.

SECONDARY OUTCOMES:
Secondary Outcome 1: Late PONV | First three postoperative days
  Incidence of postoperative nausea and vomiting within the first three postoperative days
Secondary Outcome 2: Modified Aldrete Score | First two postoperative hours
  A score to assess readiness of discharge from postanesthesia care unit (PACU). Patients can achieve 0-14 points in the modified Aldrete Score. A modified Aldrete Score > 12 points signals that criteria for discharge from PACU have been fulfilled, a modified Aldrete Score < 12 points signals that patients should stay in PACU.
Secondary Outcome 3: Ready for Hospital Discharge Scale | First three postoperative days
  A score to evaluate patients' subjective readiness for hospital discharge. Patients can achieve 0-80 points in the Ready for Hospital Discharge Scale. Higher scores mean that patients are ready for hospital discharge, lower scores mean that patients are not ready for hospital discharge.

OTHER OUTCOMES:
Exploratory Outcome 1: Intraoperative cerebral oxygen saturation between study groups | Throughout surgery
  Intraoperative non-invasive near-infrared spectroscopy for measurement of cerebral oxygenation.
Exploratory Outcome 2: Intraoperative cerebral oxygen saturation between patients, who experienced PONV, and patients without PONV | Throughout surgery and first two postoperative hours
  Intraoperative non-invasive near-infrared spectroscopy for measurement of cerebral oxygenation.
Exploratory Outcome 3: Impact of Event Scale-Revised | Before surgery
  A self-report measure to evaluate the presence of posttraumatic stress disorder. It consists of 22 items, which are rated on a 4-point scale ranging from 0 ("not at all") to 4 ("extremely"). Values are added up for the avoidance subscale, the intrusion subscale and the hyperarousal subcale and X is calculated via the following formula: X = (-0,02 x Intrusion) + (0,07 x Avoidance) + (0,15 x Hyperarousal) - 4,36. A value for X > 0 indicates the likely presence of PTSD.
Substudy 1: Preoperative Copeptin | Before surgery
  Comparison between preoperative Copeptin concentrations between patients with and without PONV.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Reiterer, MD, Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No
We will not share any individual participant data